CLINICAL TRIAL: NCT01326260
Title: Early Aggressive Correction of Severe Acidosis With Tris-hydroxymethylaminomethane (THAM) in Patients With Severe Traumatic Injury: A Retrospective Cohort Study
Brief Title: Early Aggressive Correction of Severe Acidosis With Tris-hydroxymethylaminomethane (THAM)
Acronym: THAM
Status: Terminated | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CHR 10-02652
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Resuscitation, Trauma Patients
Keywords: resuscitation; trauma; THAM; colloids; crystalloids
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- THAM Patients: Patients who were managed with the use of THAM
- Non-THAM Patients: Patients who did not use THAM but were resuscitated with crystalloids and colloids and may have received sodium bicarbonate for the treatment of acidosis

SUMMARY:
This study involved the medical record review of resuscitation records for all severely-injured trauma patients requiring emergent surgical intervention and significant acidosis from 2005 through 2009.

DETAILED DESCRIPTION:
The study objective is to assess the efficacy of fluid resuscitation and treatment of acidosis in patients who were managed with use of amine buffer THAM (tris-hydroxymethlaminomethane) versus those who were resuscitated with crystalloids or colloids and may have have received sodium bicarbonate for the treatment of acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of severe traumatic injury requiring emergent surgery
* Peri-operative development of severe acidosis (defined arterial ph less than or equal to 7.20 or base deficit greater than or equal to 10 mEq/dL)
* Acidosis was treated with either THAM or "usual care" (defined as crystalloid either or without sodium bicarbonate)

Exclusion Criteria:

* None

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to San Francisco General Hospital from 2005 through 2009 with severe traumatic injury requiring emergent surgery who develop severe acidosis
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Total amount of fluids and blood products used during the operative and 72 hr post-operative period. | Operative period and ICU (72 hr) post-op period
  Total amount of fluids and blood products used during the operative and 72 hr post-operative period.

SECONDARY OUTCOMES:
Intra-operative, intensive care unit and hospital mortality | From the operative procedure onset to discharge out of the ICU or expiration
  Measure the the number of mortality during intra-operative and/or ICU period

CONTACTS AND LOCATIONS:
Overall Officials: Julin Tang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco at San Francisco General Hospital, San Francisco, California, United States